CLINICAL TRIAL: NCT05535361
Title: A Feasibility Study to Evaluate Safety and Probable Benefit of the Eclipse XL1 System for Distraction Enterogenesis in Adult and Pediatric Patients With Short Bowel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eclipse Regenesis, Inc. (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Children's Hospital Medical Center, Cincinnati (Other); Stanford University (Other); University of California, San Francisco (Other); Boston Children's Hospital (Other); Lucile Packard Children's Hospital at Stanford (Unknown); Children's National Health System, Washington DC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0001; R44DK127658 (NIH)
Record Dates: First submitted 2022-09-01; First posted 2022-09-10 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Short Bowel Syndrome
Keywords: short bowel syndrome; intestinal failure; Necrotizing enterocolitis; short gut; intestinal volvulus; intestinal atresia
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Failure; Enterocolitis, Necrotizing; Intestinal Volvulus; Intestinal Atresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Eclipse XL1 Coil Treatment Group (Experimental): All subjects will be assigned to the XL1 Coil treatment group.
  Interventions: Device: Distraction Enterogenesis in Adult Patients with Short Bowel Syndrome

INTERVENTIONS:
Device: Distraction Enterogenesis in Adult Patients with Short Bowel Syndrome — The surgeon verifies the intestinal diameter and selects the appropriate device diameter size. The device is introduced into the lumen of the intestine and advanced about 5-10cm. The surgeon uses 4-0 chromic sutures placed in the seromuscular layer to secure the XL1 Coil within the intestine. The surgeon places metal clips on proximal and distal sutures and in the mesentery adjacent to the XL1 Coil ends to mark the location for radiologic evaluation. The surgeon releases the XL1 Coil and closes the enterotomy.

SUMMARY:
A Feasibility Study to Evaluate Safety and Probable Benefit of the Eclipse XL1 System for Distraction Enterogenesis in Adult and Pediatric Patients with Short Bowel Syndrome

DETAILED DESCRIPTION:
This clinical investigation is a study to evaluate safety and probable benefit of the Eclipse XL1 System in pediatric and adult subjects with short bowel syndrome. This study is a single arm study and will enroll subjects ages 3 months to 65 years old at up to 10 study sites in the United States. This study will be open label; treatment allocation will be known by the subjects, the Principal Investigator and his medical staff. Recruitment is expected to occur over the course of 24-36 months.

Device placement will be administered during a standalone procedure or a previously planned procedure that is otherwise needed by the study subject. Subjects may receive up to 2 devices at one time and/or have multiple procedures over time based on clinical necessity Study objectives will be monitored by reviewing patient nutrition, weight, and stool assessment data. The study device will also monitored by radiographic examination to confirm location of the device and assess the safety and probable benefit of distraction enterogenesis until the device is removed or passes out of the intestine naturally. Patients will be followed while the study device is in situ and at 3 and 6 months post device passing or removal. Subjects may or may not be discharged from the hospital while participating in the study, and investigators may recommend that a subject stay in-patient for a portion or the entire length of study, depending on subject health.

ELIGIBILITY:
Inclusion Criteria:

* Subject has short bowel syndrome, defined as 50% or less of expected bowel length based on subject age and/or height, and measured at the time of the subject's prior intestinal resection.
* Minimum residual bowel length of 3 cm.
* Male or female patients aged 3 mo to 65 years inclusive
* The subject, parent or legal guardian of the subject is able to read, understand, and is willing to provide informed consent.
* The subject or parent or legal guardian of the patient is able to understand the requirements of the study and is willing to bring the subject to all clinic visits and complete all study related procedures (as determined by the investigator).

Exclusion Criteria:

* Ultra-short bowel syndrome defined as less than 3 cm of bowel length.
* Diagnosed Inflammatory bowel disease-unclassified (not Crohn's or ulcerative colitis)
* Evidence of active or prior Crohn's disease.
* Primary intestinal failure (i.e., without loss or resection of intestinal tissue).
* Coagulopathy, as defined by INR > 1.4 or platelets < 100.
* Known immunocompromised status including, but not limited to, individuals who have undergone organ transplantation, chemotherapy or radiotherapy within the past 12 months, who have clinically significant leukopenia, who are positive for the human immunodeficiency virus (HIV) or whose immune status makes the subject a poor candidate for clinical trial participation in the opinion of the Investigator.
* Subject is determined by the investigator to be unsuitable for participation in this trial for any reason.

Ages: 3 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Device and procedure related adverse events | 4 to 6 months
  Incident rate of moderate or severe procedure and/or device related adverse events

SECONDARY OUTCOMES:
Assess the lengthening of the small intestine | 4 to 6 months
  Assess the lengthening of the small intestine via the Eclipse XL1 Coil.
Improvement in overall nutritional status | 6 to 12 months
  Improvement in overall nutritional status at 6 months post final implantation compared to pre-procedure as evidenced by change in parenteral, enteral, oral intake; stool frequency and quality; weight.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park J, Puapong DP, Wu BM, Atkinson JB, Dunn JC. Enterogenesis by mechanical lengthening: morphology and function of the lengthened small intestine. J Pediatr Surg. 2004 Dec;39(12):1823-7. doi: 10.1016/j.jpedsurg.2004.08.022. PMID 15616941
- [Background] Chang PC, Mendoza J, Park J, Lam MM, Wu B, Atkinson JB, Dunn JC. Sustainability of mechanically lengthened bowel in rats. J Pediatr Surg. 2006 Dec;41(12):2019-22. doi: 10.1016/j.jpedsurg.2006.08.014. PMID 17161196
- [Background] Mendoza J, Chang CY, Blalock CL, Atkinson JB, Wu BM, Dunn JC. Contractile function of the mechanically lengthened intestine. J Surg Res. 2006 Nov;136(1):8-12. doi: 10.1016/j.jss.2006.01.027. Epub 2006 Sep 18. PMID 16979663
- [Background] Shekherdimian S, Scott A, Chan A, Dunn JC. Intestinal lengthening in rats after massive small intestinal resection. Surgery. 2009 Aug;146(2):291-5. doi: 10.1016/j.surg.2009.03.034. Epub 2009 Jun 21. PMID 19628087